CLINICAL TRIAL: NCT04917120
Title: Observational Prospective Study Measuring the Impact of the Use of a Hypnotic Script Associated With Virtual Reality on the Pain of the Child's Sickle Cell During a Vaso-occlusive Crisis
Acronym: DREPAReV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: APHP201280; IDRCB2020-AO2248-31 (Other: ANSM)
Record Dates: First submitted 2021-05-10; First posted 2021-06-08 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-05

CONDITIONS: Sickle Cell Disease
Keywords: Sickle cell disease; Pain; Virtual reality; Vaso occlusive crises; Hypnosis
MeSH Terms: conditions — Anemia, Sickle Cell; Pain; Vaso-Occlusive Crises

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- VRH (virtual reality hypnosis) (Experimental)
  Interventions: Device: Virtual Reality

INTERVENTIONS:
Device: Virtual Reality — The procedure will consist of a virtual reality program associated with suggestions of hypnoanalgesia, be added to usual care. Included patients will benefit from the Virtual Reality program combined with hypnoanalgesia suggestions for a period of 20 minutes. We will use a helmet with a built-in screen and an audio headset connected to a control room. Patients will watch an Virtual Reality sequence while listening to narratives designed for the hypnoanalgesia of the present pain.

SUMMARY:
The purpose of this study is to evaluate the effect of Virtual Reality induced Hypnosis on patients' pain scores, anxiety and the use of analgesics during a vaso-occlusive crisis

DETAILED DESCRIPTION:
Virtual reality hypnosis could probably reduce vaso-occlusive crisis-related (vaso-occlusive crisis) anxiety and pain and provide the patient with means of optimizing the ability to cope with the painful and anxiety-provoking situations encountered in general pediatric unit.

However, this non-pharmacological analgesic technique is little used in the context of vaso-occlusive crisis in children and adolescents in French pediatric services.

Currently, the average pain scores of children and adolescents hospitalized for vaso-occlusive crisis after treatment in the emergency department is 6 out of 10 on a simple numerical scale (according to a preliminary study conducted on 30 files of sickle cell disease patients over 6 years of age hospitalized in general pediatrics, Trousseau AP-HP hospital over a period of 6 months in 2018), despite the implementation of optimal pharmacological means with regard to the HAS analgesia recommendations. The pain score stays high despite a well-conducted analgesic treatment.

Our hypothesis is that virtual reality hypnosis could potentiate the effects of virtual reality by hypnotic suggestions specific to the pain of patients with vaso-occlusive crisis . This is a pain and anxiety reduction strategy that has, to our knowledge, never been evaluated.

So this is innovative by the method but also of the pediatric target population suffering from recurrent and severe pain.

A session of hypnoanalgesia suggestions associated with a virtual reality program will allow the patient to acquire the necessary competence to manage with his or her pain and thus be more autonomous in its management.

The physiopathological hypothesis of the research is that the immersion of the patient with vaso-occlusive crises related pain during a hypnotic experience induced by virtual reality allows to saturate his sensoriality, thus reducing nociceptive perceptions and vaso-occlusive crisis -related anxiety. We hypothesize that this experiment is feasible and that it can produce decrease in pain and anxiety scores for children benefiting from a virtual reality hypnosis session during vaso-occlusive crisis within one hour of session.

ELIGIBILITY:
Inclusion Criteria:

* Child over 6 years of age on the day of acceptance of the study (no upper limit)
* Suffering from sickle cell disease whatever genotype
* Admission in hospital for a VOC (vaso-occlusive crisis)
* Informed and signed consent by at least one legal guardian, if child is minor, and verbal agreement of the child himself.

Exclusion Criteria:

* Deaf patient, visually impaired patient, claustrophobic and/or aquaphobic patient
* Patient not understanding French
* History of psychiatric illness such as paranoia, schizophrenia, manic-depressive psychosis, high suicide risk patient.

The patient may be included several times in the study if he is hospitalized again during the inclusion period.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Actual)
Dates: Start 2021-07-13 (Actual); Primary Completion 2022-07-19 (Actual); Study Completion 2022-07-19 (Actual)

PRIMARY OUTCOMES:
pain assessment with score (patient) | hours 3 after a virtual reality
  Measuring pain thanks to score pain by the patient 3 hours after a Virtual Reality session performed within the first 6 hours after arrival in the general pediatrics unit Patients will use le Faces Pain Scale - Revised.

SECONDARY OUTCOMES:
pain assessment with score (patient) | 10 minutes before HVR
  Measuring pain thanks to score pain by the patient 10 minutes before the Virtual Reality session performed within the first 6 hours after arrival in the general pediatrics unit Patients will use le Faces Pain Scale - Revised.
pain assessment with score (patient) | 1 hour after a virtual reality
  Measuring pain thanks to score pain by the patient 1 hour after a Virtual Reality session performed within the first 6 hours after arrival in the general pediatrics unit Patients will use le Faces Pain Scale - Revised.
pain assessment with score (health care personnel) | 10 minutes before HVR
  Measuring pain thanks to score pain by the health care personnel 10 minutes before the Virtual Reality session performed within the first 6 hours after arrival in the general pediatrics unit Health care personnel will use EVENDOL score (score between " 0 " corresponding to " no pain sign " and " 15 " corresponding to " maximum pain signs ").
pain assessment with score (health care personnel) | 1 hour after a virtual reality
  Measuring pain thanks to score pain by the health care personnel 1 hour after a Virtual Reality session performed within the first 6 hours after arrival in the general pediatrics unit Health care personnel will use EVENDOL score (score between " 0 " corresponding to " no pain sign " and " 15 " corresponding to " maximum pain signs ").
pain assessment with score (health care personnel) | 3 hour after a virtual reality
  Measuring pain thanks to score pain by the health care personnel 3 hours after a Virtual Reality session performed within the first 6 hours after arrival in the general pediatrics unit Health care personnel will use EVENDOL score (score between " 0 " corresponding to " no pain sign " and " 15 " corresponding to " maximum pain signs ").
anxiety assessment | 10 minutes before HVR
  To assess efficacy on anxiety 10 minutes before the session, we will use a numerical scale graduated from 0 to 10 (" 0 " corresponding to " no anxiety " and " 10 " corresponding to " maximum anxiety ")
anxiety assessment | 1 hour after HVR
  To assess efficacy on anxiety 1 hour after the session, we will use a numerical scale graduated from 0 to 10 (" 0 " corresponding to " no anxiety " and " 10 " corresponding to " maximum anxiety ")
anxiety assessment | 3 hour after HVR
  To assess efficacy on anxiety 3 hours after the session, we will use a numerical scale graduated from 0 to 10 (" 0 " corresponding to " no anxiety " and " 10 " corresponding to " maximum anxiety ")
patient satisfaction assessment | 3 hour
  We will use the Likert scale 3 hours after the session (" 0 " corresponding to " no satisfaction " and " 5 " corresponding to " complete satisfaction "
health care personnel satisfaction assessment | 5 months
  We will use the Likert scale 3 hours after the session (" 0 " corresponding to " no satisfaction " and " 5 " corresponding to " complete satisfaction "

CONTACTS AND LOCATIONS:
Overall Officials: Sophie DUGUE, Study Chair — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Trousseau Hospital, General pediatric departement, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided